CLINICAL TRIAL: NCT05153278
Title: Effectiveness and Impact of Intravenous Iron Versus Standard Treatment in Treating Iron Deficiency Anemia in the Emergency Department at University Medical Center
Brief Title: IV Iron Versus Standard Treatment for Iron Deficiency Anemia in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Gregory Patek, MD, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E18152
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia Treatment; Iron-deficiency; Iron Deficiency Anemia Due to Blood Loss; Iron Deficiency Anemia
Keywords: iron deficiency anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Infusion Pumps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: Patients that received standard treatment (packed red blood cells) for iron deficiency anemia
  Interventions: Biological: Packed red blood cells
- Experimental group: Patients that received intravenous iron instead of standard treatment (packed red blood cells) for iron deficiency anemia
  Interventions: Drug: Intravenous drug

INTERVENTIONS:
Biological: Packed red blood cells — Standard treatment for iron deficiency anemia (control)
  Other Names: PRBC
  Groups: Control group
Drug: Intravenous drug — Experimental treatment for iron deficiency treatment
  Other Names: Intravenous iron
  Groups: Experimental group

SUMMARY:
The investigators will retrospectively collect data of patients infused at UMC's emergency department (ED) with long acting irons (ferric carboxymaltose, iron dextran, iron sucrose, etc.), in addition, patients infused with blood products, with intent to treat iron deficiency anemia (IDA). Patient records reviewed will be from patients who were infused at UMC ED from January 2013 to June 2018. Primary aim of analysis will be to investigate superiority between interventions implemented for treating IDA. In addition, the investigators will utilize data to characterize patients who used ED services as an avenue to receive treatment for IDA. Further, the investigators will conduct cost analysis between different IDA directed treatments administered in the ED at UMC.

DETAILED DESCRIPTION:
Background:

Iron deficiency anemia (IDA) is a condition that impacts approximately 2-billion people globally, and impacts individuals from all socioeconomic backgrounds, making it one of the most common nutritional disorders in the world. In any population, women and children are the groups that are more susceptible to suffering from IDA [3]. IDA has broad influences on the health of an individual, ranging from cognitive decline to motor deficits. When coupled with pregnancy, IDA has been shown to be associated with low birth weight and carries an increased risk of maternal and perinatal mortality. In addition to women and children, the prevalence of IDA has been found to increase with age, and with chronic disease. The approach to treating IDA regularly begins with oral iron supplementation. However, due to increased gastrointestinal side effects or excessive losses of iron, intravenous iron has been shown to be better tolerated. Further, intravenous iron is another attractable iron replacement strategy in IDA when the need for rapid delivery is required, such as in pregnancy or following traumas. When compared to blood products, intravenous iron is an attractive option due to its ready availability. With a growing and aging population it is important that major health problems such as IDA be investigated further in order to identify sustainable therapeutic strategies.

Benefits of Study:

This retrospective study will provide the investigators with valuable knowledge on which treatment for IDA may be most effective in treating our El Paso population of patients suffering from IDA (Primary Aim). This study will also allow the investigators to identify which IDA treatment is most cost effective (Secondary Aim A), and which population of the community would benefit the most from an outpatient infusion service (Secondary Aim B).

Chart Inclusion Criteria:

All patients receiving one IDA intervention in the UMC ED who had at least one complete blood count or hemoglobin after discharge from the emergency department or hospital.

Exclusion Criteria:

Patients with no records of follow up.

Identification:

Collection of Patient Records and Data: Patient records reviewed will be from patients who were infused at UMC ED from January 2013 to June 2018. The age group of patients will be those greater than 18 years of age. The investigators will include all patients presenting to or treated at UMC ED during this five and one-half year period. Patient information such as unique identifiers (e.g. medical record number, hospital account number) will be used to navigate patient records for approved research personnel only. No procedures will be performed as part of this study. All data will be collected as a retrospective chart review. The investigators will access patient data through both UMC and Texas Tech electronic medical records as patients who received an intervention may have received follow up in a Texas Tech clinic rather than the UMC emergency department. The only risk of this study is the potential for loss of confidentiality. Research personnel will take extra measures to reduce this risk. The researchers will not publish any data that can be used to identify the patient, such as but not limited to personal or unique identifiers, medical record numbers, hospital account numbers or date of birth.

Experiment group:

Patient charts will be identified through digital records of UMC pharmacy and UMC blood bank. Patients included, will be those listed to have IDA by set criteria [Listed below], and who were treated with at least one IDA intervention other than blood product transfusion. Control group will be formed using patients who received at least one IDA intervention using blood product transfusion only. The investigators will attempt to match charts by age, condition leading to IDA, and gender in final analysis.

Set criteria:

Patient charts will be identified if they were the recipient of listed blood and bloodless transfusion products for treatment of IDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving one IDA intervention in the UMC ED who had at least one complete blood count or hemoglobin after discharge from the emergency department or hospital

Exclusion Criteria:

* Patients with no records of follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iron deficiency anemia treated with intravenous iron or packed red blood cells
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin | 180 days
  Change in serum hemoglobin over time

SECONDARY OUTCOMES:
Change in MCV (mean corpuscular volume) | 180 days
  Change in MCV over time

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Patek, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University Health Sciences Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No